CLINICAL TRIAL: NCT00257387
Title: A Nonrandomized, Open-label, Multicenter, Sequential Phase Study to Evaluate the Safety and Efficacy of Cyclosporine Dose Reduction and Cyclosporine Elimination in Chinese De Novo Renal Allograft Recipients Receiving Rapamune
Brief Title: Study Evaluating Cyclosporine Dose Reduction and Cyclosporine Elimination in Chinese Kidney Transplants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0468H1-101308
Record Dates: First submitted 2005-11-04; First posted 2005-11-22 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2007-06

CONDITIONS: Kidney Transplant
Keywords: Kidney; Kidney Transplant
MeSH Terms: interventions — Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine

SUMMARY:
Evaluate the incidence of acute rejection at 12 months after transplantation in subjects receiving induction therapy with cyclosporine microemulsion (CsA) and Rapamune followed by CsA dose reduction (Phase I) with subjects receiving induction therapy with CsA and Rapamune followed by CsA discontinuation (Phase II) in Chinese de novo renal allograft recipients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end-stage renal disease scheduled to receive a primary renal allograft from a cadaveric donor, from a living-unrelated donor, or a living-related HLA-mismatched donor.
* Subjects must be at least 18 years of age.

Exclusion Criteria:

* Subjects with active major infection, including active hepatitis B or C infection, HIV, decreased platelets, elevated lipids, or multiple organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of acute rejection in renal allograft recipients at 6 months post-transplantation.

SECONDARY OUTCOMES:
To evaluate the treatment groups with respect to incidence of adverse events, renal function, subject and graft survival at 6 and 12 months, and the incidence and severity of acute rejection at 12 months post-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer